CLINICAL TRIAL: NCT02911480
Title: Assessment of Pharmacokinetics and Bioavailability of Carbon-14 ([14C])-Labelled Oxytocin
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Study/financial issues
Sponsor: Oxytone Bioscience BV (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: OXB-001
Record Dates: First submitted 2016-09-16; First posted 2016-09-22 (Estimated); Last update posted 2018-04-06 (Actual); Status verified 2018-04

CONDITIONS: Healthy Women of Child Bearing Potential
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- oxytocin intravenous 0.1 IU (Experimental): single dose of 0.1 International Units (IU) intravenous (IV) oxytocin
  Interventions: Drug: Oxytocin
- oxytocin intravenous 1 IU (Experimental): single dose of 1 IU IV oxytocin
  Interventions: Drug: Oxytocin
- oxytocin intravenous 10 IU (Experimental): single dose of 10 IU IV oxytocin
  Interventions: Drug: Oxytocin
- oxytocin tablet 20 IU (Experimental): single dose of 20 IU tablet oxytocin
  Interventions: Drug: Oxytocin
- oxytocin tablet 200 IU (Experimental): single dose of 200 IU tablet oxytocin
  Interventions: Drug: Oxytocin

INTERVENTIONS:
Drug: Oxytocin

SUMMARY:
The current study is designed as a phase I multiple dose study to evaluate the pharmacokinetics and bioavailability of [14C]-labelled oxytocin in healthy women.

ELIGIBILITY:
Inclusion Criteria:

* Non-smoking women of child bearing potential (WOCBP)
* Body mass index (BMI) between ≥ 18.0 and ≤ 30.0 kg/m2
* Subject must voluntarily sign a written informed consent agreement approved by the Independent Ethics Committee (IEC) after explanation of the nature and objectives of the study and before any study specific procedure
* Subject must be in good physical and mental health as judged by the Investigator based on evaluation of medical and gynecological history, physical examination, clinical laboratory, ECG, and vital signs data
* Subject is willing and able to comply with all conditions and requirements of the study

Exclusion Criteria:

* Lactation and/or pregnancy in the previous 6 months before screening, whichever is applicable
* Intention to become pregnant during the study or within 1 months after the follow up visit
* History of, or existing thromboembolic, cardiovascular or cerebrovascular disorder
* Treatment for any major psychiatric disorder in the previous 12 months or use of antidepressant medication before screening
* Any clinically significant abnormality following review of medical history, laboratory results and physical examination at screening as judged by the Investigator
* Conditions or disorders that might affect the absorption, distribution, metabolism or excretion of the study drugs
* Contraindications for the use of oxytocin
* Hypersensitivity to the active substances or to any of the excipients of the investigational product or reference therapy
* Present use or use within 30 days before the start of the study medication of one or more of the following medications: antihypertensive drugs, anti-coagulant therapy, medication that could affect myometrial contractility, sex steroids, prostaglandins and its analogues, inhalation anesthetics, vasoconstrictors/sympathomimetics and caudal anesthetics, vasopressin-like drugs
* Use of any prescribed or over-the-counter medication within 14 days before Day 1
* Administration of any other investigational drug within 3 months before Day 1 or participation in 3 or more clinical trials in the 10 months before Day 1
* Loss of more than 500 milliliters (mL) blood during the 3 months before Day 1, or intention to donate blood in the 3 months after completing the study
* Subjects with a positive test result for hepatitis B, hepatitis C, or human immunodeficiency virus (HIV) at screening
* Subjects with a history of alcohol or drug abuse or with a positive result at screening, for tests of alcohol intake or drugs of abuse

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Estimated); Primary Completion 2017-02 (Estimated); Study Completion 2017-08-31 (Actual)

PRIMARY OUTCOMES:
pharmacokinetics (PK) parameter for oxytocin: maximum plasma concentration (Cmax) | Day 1, predose and at t=3, 7, 10, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, 360, 480 minutes.
pharmacokinetics (PK) parameter for oxytocin: time to Cmax (tmax) | Day 1, predose and at t=3, 7, 10, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, 360, 480 minutes.
pharmacokinetics (PK) parameter for oxytocin: area under the plasma-concentration time curve (AUC) | Day 1, predose and at t=3, 7, 10, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, 360, 480 minutes.
pharmacokinetics (PK) parameter for oxytocin: terminal half-life (t1/2) | Day 1, predose and at t=3, 7, 10, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, 360, 480 minutes.
pharmacokinetics (PK) parameter for oxytocin: bioavailability (F) | Day 1, predose and at t=3, 7, 10, 20, 30, 45, 60, 90, 120, 150, 180, 240, 300, 360, 480 minutes.